CLINICAL TRIAL: NCT04821089
Title: A Phase Ib/II, Multicentre, Double-blind, Randomised, Placebo-controlled, Dose Escalation and Dose-finding Study to Evaluate the Safety and Efficacy of IPN10200 in Improving the Appearance of Moderate to Severe Upper Facial Lines in Adults
Brief Title: A Study to Assess the Safety and Efficacy of IPN10200 in Adult Participants With Moderate to Severe Upper Facial Lines
Acronym: LANTIC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-FR-10200-002; 2024-512782-14-00 (EU CTIS Number)
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Moderate to Severe Upper Facial Lines
MeSH Terms: interventions — abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IPN10200 group (Experimental): Stage 1/Step 1: Several cohorts of participants will be randomized in a ratio of 3:1 in a dose-escalation manner. The decision to escalate to the next dose for each cohort will be based on Data Monitoring Committee (DMC) recommendation.
  Stage 1/Step 2: parallel dose-ranging manner Stage 1/Step 3: each cohort will include three treatment groups randomised in a ratio of 4:1:1 The decision to escalate to the next dose for each cohort will be based on DMC recommendation .
  Stage 2: the dose(s) chosen for administration in each region of the face will be selected on the basis of the intermediate analyses of Stage 1/Step 3. Participants will be randomised for each group in a ratio of 4:4:1.
  Stage 3: total dose for each region defined in Stages 1 and 2. Participants will be randomised for each group in a ratio of 3:1.
  Interventions: Biological: IPN10200
- Placebo group (Placebo Comparator): Stage 1/Step 1: Several cohorts of participants will be randomized in a ratio of 3:1 in a dose-escalation manner. The decision to escalate to the next dose for each cohort will be based on Data Monitoring Committee (DMC) recommendation.
  Stage 1/Step 2: parallel dose-ranging manner Stage 1/Step 3: each cohort will include three treatment groups randomised in a ratio of 4:1:1 The decision to escalate to the next dose for each cohort will be based on DMC recommendation.
  Stage 2: the dose(s) chosen for administration in each region of the face will be selected on the basis of the intermediate analyses of Stage 1/Step 3. Participants will be randomised for each group in a ratio of 4:4:1.
  Stage 3: total dose for each region defined in Stages 1 and 2. Participants will be randomised for each group in a ratio of 3:1.
  Interventions: Biological: IPN10200 Placebo
- Dysport group (stage 1 / step 2 and 3 only) (Active Comparator)
  Interventions: Biological: Dysport

INTERVENTIONS:
Biological: IPN10200 — Stage 1: Several different doses will be administrated in a dose-escalation manner.
  One single injection will be injected locally into several sites across the glabellar region.
  Stage 2: One single injection will be injected locally into several sites across the glabellar, forehead and lateral Canthal regions.
  Stage 3: One single injection will be injected locally into several sites across the upper facial area.
  Arms: IPN10200 group
Biological: IPN10200 Placebo — Stage 1: One single injection of study intervention will be injected locally into several sites across the glabellar region.
  Stage 2: One single injection will be injected locally into several sites across the glabellar, forehead and lateral Canthal regions.
  Stage 3: One single injection will be injected locally into several sites across the upper facial area.
  Arms: Placebo group
Biological: Dysport — Single administration of study intervention in stage 1 / step 2 and 3 only
  Arms: Dysport group (stage 1 / step 2 and 3 only)

SUMMARY:
The purpose of this study is to assess the safety and efficacy profile of increasing doses of IPN10200 in comparison to placebo, with the aim to discover the doses(s) that offer the best efficacy/safety profile when used for the treatment of moderate to severe Upper Facial Lines.

This study will be conducted in three stages. The full study (including all stages) will have a maximum 727 participants.

Stage 1 (phase Ib & II)

* Step 1 (Phase Ib): a dose-escalation first-in-human step in participants with moderate to severe Glabellar Lines (GL)
* Step 2 (Phase II): dose ranging step in participants with moderate to severe GL as compared with Dysport
* Step 3 (Phase II): dose finding step in participants with moderate to severe GL as compared with Dysport, followed by an open label (OL) phase for the highest dose cohort to assess the long-term safety and efficacy of IPN10200. In the OL phase, participants may receive repeat administrations of IPN10200 for up to three additional cycles (up to four treatment cycles in total during the study).

Stage 2 (phase II) - An evaluation of efficacy and safety of IPN10200 in one of the following regions: GL + forehead lines (FHL), forehead lines (FHL) or lateral canthal lines (LCL)

Stage 3 (phase II)

- A safety and efficacy evaluation of IPN10200 in all three regions (GL, FHL and LCL)

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
2. Moderate or severe (Grade 2 or 3) GL (Stage 1) at maximum contraction at Baseline, as assessed by the ILA using a validated 4-point photographic scale.
3. Moderate or severe (Grade 2 or 3) GL (Stage 1) at maximum contraction at Baseline, as assessed by the SSA using a validated 4-point categorical scale.
4. Moderate or severe (Grade 2 or 3) FHL (Stage 2) at maximum contraction and moderate to severe GL at maximum contraction at Baseline or moderate to severe (Grade 2 or 3) LCL (Stage 2) at maximum contraction (Stage as assessed by the ILA using a 4-point photographic scale).
5. Moderate or severe (Grade 2 or 3) FHL (Stage 3) at maximum contraction and moderate to severe GL at maximum contraction at Baseline and moderate to severe (Grade 2 or 3) LCL (Stage 3) at maximum contraction (Stage as assessed by the ILA using a 4-point photographic scale).
6. Moderate or severe (Grade 2 or 3) FHL (Stage 2) at maximum contraction and moderate to severe GL maximum contraction at Baseline or moderate to severe (Grade 2 or 3) LCL (Stage 2) at maximum contraction as assessed by the SSA using a 4-point photographic scale.
7. Moderate or severe (Grade 2 or 3) FHL (Stage 3) at maximum contraction and moderate to severe GL maximum contraction at Baseline and moderate to severe (Grade 2 or 3) LCL (Stage 3) at maximum contraction, as assessed by the SSA using a 4-point photographic scale.
8. Dissatisfied or very dissatisfied (Grade 2 or 3) with their lines (Stages 1 to 3) at Baseline, as assessed by the SLS.
9. Male and female participants (only female for Stage 1/Step 1). Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
10. Capable of giving signed informed consent includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
11. Participant has both the time and the ability to complete the study and comply with study instructions.
12. Does not reside in an institution by administrative or court order.
13. Is not a sponsor employee or clinical research unit personnel directly affiliated with the study or is not an immediate family member. Immediate family is defined as a spouse, parent, child or sibling whether biological or legally adopted.

Exclusion Criteria:

1. An active infection or other skin problems in the upper face including the GL, FHL, and LCL area (e.g. acute acne lesions or ulcers).
2. A history of eyelid blepharoplasty or brow lift within the past 5 years
3. A history of facial nerve palsy.
4. Marked facial asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin.
5. Any known medical condition that may put the participant at increased risk in regard to exposure to BoNT of any serotype (i.e. myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, etc.)
6. Has COVID-19 illness or a known positive SARS-CoV-2 test (Stage 1), or the presence of any other condition (e.g. neuromuscular disorder or other disorder that could interfere with neuromuscular function)
7. Previous treatment with any BoNT serotype for Stage 1 / Step 1 or any recent treatment (within the past 9 months prior to baseline) with any BoNT serotype for Stage 1 / Step 2, Stage 1/Step 3, Stages 2 and 3. Participants treated in earlier Stages/Steps of the study must not be included in any later Stages/Steps.
8. Any prior treatment with permanent fillers in the upper face including the GL, FHL and LCL area.
9. Any prior treatment with long lasting dermal fillers or any permanent procedures in the upper face inclusion the GL area within the past 3 years and/or skin abrasions/resurfacing (whatever the interventional technic used) within the past 5 years, or photo rejuvenation or skin/vascular laser intervention within the 12 months prior to Baseline.
10. Any planned facial cosmetic surgery during the study.
11. Use of concomitant therapy which, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study intervention. Therapy considered necessary for the participant's welfare may be given at the discretion of the investigator.
12. Use of medications that affect neuromuscular transmission, such as curare-like non depolarising agents, lincosamides, polymyxins, anticholinesterases, aminoglycoside antibiotics and systemic retinoids, within the past 30 days prior to Baseline.
13. Use of any experimental device within 30 days or use of any treatment with an experimental drug within five times the documented terminal half-life of the respective drug or its metabolites or if the halflife is unknown within 30 days prior to the start of the study (prior to Baseline) and during the conduct of the study.
14. Known positive for hepatitis B antigen, or hepatitis C virus antibody, or for human immunodeficiency virus (HIV) or a diagnosis of acquired immunodeficiency syndrome.
15. Clinically diagnosed significant anxiety disorder, or any other significant psychiatric disorder (e.g. depression) that might interfere with the participant's participation in the study
16. An inability to substantially lessen GL and/or horizontal forehead rhytids even by physically spreading them apart as determined by the investigator.
17. Known allergy or hypersensitivity to BoNT or any excipients of IPN10200 or Dusport/Azzalure, or allergy to cow's milk protein.
18. A history of drug or alcohol abuse
19. Pregnant women, nursing women, premenopausal women or women of childbearing potential not willing to practice a highly effective form of contraception method
20. Male participants who are not vasectomized and who have female partners of childbearing potential and are not willing to use condoms with spermicide throughout study participation.
21. Any uncontrolled systemic disease or other significant medical condition which would be harmful for the participant to be entered into the study or continue participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 727 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) at each dose | From the baseline to the end of the study (9 months)
  At Stage 1/Step 1, Stage 3
Incidence of serious adverse events (SAEs) at each dose | From the baseline to the end of the study (9 months)
  At Stage 1/Step 1, Stage 3
Incidence of Adverse Events (AEs) (or SAEs) leading to withdrawals and Adverse Events of Special Interest (AESIs) | From the baseline to the end of the study (9 months)
  At Stage 1/Step 1, Stage 3
Response to treatment as measured by the composite response of 2-grade improvement on Investigator's Live Assessment (ILA) at maximum contraction | At Week 4
  At stage 1/Step 2, Step 3; ILA: a validated 4-point photographic scale to assess the severity and appearance of the GLs at maximum frown and at rest where 0 is "no lines are noticeable" and 3 is "lines are extremely pronounced"
Response to treatment as measured by the composite response of 2-grade improvement on subject's self-assessment (SSA) at maximum contraction | At Week 4
  At Stage 1/Step 2 and Step 3; SSA: a validated 4-point categorical scale to assess the appearance of their Glabellar Lines (GLs) at maximum frown where 0 is "no wrinkles" and 3 is "severe wrinkles".
Response to treatment as measured by the composite response of 2-grade improvement on ILA at maximum contraction on the forehead lines (FHL) area | At Week 4
  At Stage 2 for the glabellar lines (GL)+ FHL group
Response to treatment as measured by the composite response of 2-grade improvement on SSA at maximum contraction on the forehead lines (FHL) area | At Week 4
  At Stage 2 for the glabellar lines (GL)+ FHL group
Response to treatment as measured by the composite response of 2-grade improvement ILA at maximum contraction on the lateral canthal lines (LCL) area | At Week 4
  At stage 2 for the LCL group
Response to treatment as measured by the composite response of 2-grade improvement on SSA at maximum contraction on the LCL area | At Week 4
  At stage 2 for the LCL group

SECONDARY OUTCOMES:
Response to treatment measured by the composite response of 2-grade improvement on ILA | From the baseline to the end of the study (9 months)
  For all stages. ILA: a validated 4-point photographic scale to assess the severity and appearance of the GLs at maximum frown and at rest where 0 is "no lines are noticeable" and 3 is "lines are extremely pronounced"
Response to treatment measured by the composite response of 2-grade improvement on SSA | From the baseline to the end of the study (9 months)
  For all stages. SSA: a validated 4-point categorical scale to assess the appearance of their Glabellar Lines (GLs) at maximum frown where 0 is "no wrinkles" and 3 is "severe wrinkles".
Response to treatment as measured by the reduction of ≥2 grades on the ILA at maximum contraction | From the baseline to the end of the study (9 months)
Response to treatment as achieved by a score of "none" or "mild" as measured by the ILA at maximum contraction | From the baseline to the end of the study (9 months)
Response to treatment as achieved by a score of "none" or "mild" as measured by the ILA at rest | From the baseline to the end of the study (9 months)
Response to treatment as measured by the reduction of ≥2 grades on the SSA at maximum contraction | From the baseline to the end of the study (9 months)
Response to treatment as achieved by a score of "none" or "mild" as measured by the SSA at maximum contraction | From the baseline to the end of the study (9 months)
Response to treatment as achieved by a score of "very satisfied" or "satisfied" on the Subject Level of Satisfaction (SLS) | From the baseline to the end of the study (9 months)
Duration of treatment response based on ILA and SSA at maximum contraction | From the baseline to the end of the study (9 months)
Time to onset of treatment response based on subject diary cards to evaluate the appearance of their lines | From the baseline to the end of the study (9 months)
Satisfaction with facial appearance scale score on the Face-Q satisfaction scale | From the baseline to the end of the study (9 months)
  Face Q is a participant-reported outcome instrument to evaluate the experience and outcomes of aesthetic facial procedures from the participant's perspective. The Face Q is composed of over 40 scales, covering four domains (Satisfaction with Facial Appearance, Health Related Quality of Life, Adverse Effects, and Process of Care).
Incidence, severity and nature of treatment emergent adverse events (TEAEs) | From baseline to the end of the study (9 months)
Incidence, severity and nature of serious adverse events (SAEs) | From baseline to the end of the study (9 months)
Incidence, severity and nature of Adverse Events (AEs) (or SAEs) leading to withdrawals and Adverse Events of Special Interest (AESIs) | From baseline to the end of the study (9 months)
Presence of IPN10200 antibodies and titres (binding and neutralizing) | At Week 4 , Week 24 and Week 36
Presence of BoNT-A antibodies and titres (binding and neutralizing) | At Week 4 , Week 24 and Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (9):
- France (3):
  - MEDITI - Clinique Del Mar, Antibes
  - Aimed S.A.S, Lyon
  - Clinique de Chirurgie Esthétique Iéna, Paris
- Germany (6):
  - CRS Clinical Research Services Berlin GMBH, Berlin
  - Interdisciplinary Study Association, Berlin
  - ROSENPARK RESEARCH GmbH, Darmstadt
  - Privatpraxis Dr. Hilton & Partner, Düsseldorf
  - Fachbereich Chemie Institut für Biologie und Molekularbiologie Studiengang Kosmetikwissenschaft, Hamburg
  - Dermatologische Gemeinschaftspraxis Blankenfelde-Mahlow, Mahlow

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/